CLINICAL TRIAL: NCT03358069
Title: Does Emergence Time Relate With Emergence Agitation in Pediatric Patients?
Status: Completed | Type: Observational
Sponsor: Prince of Songkla University (Other)
Responsible Party: Principal Investigator, Ngamjit Pattaravit, Asst. Prof., Prince of Songkla University
Other Study IDs: PSU EA 3
Record Dates: First submitted 2017-11-02; First posted 2017-11-30 (Actual); Last update posted 2017-11-30 (Actual); Status verified 2017-11

CONDITIONS: Emergence Agitation, Post Operative Behavioral Changes
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- deep anesthetic state: technique of Anesthesia at the time of airway device removal
  Interventions: Diagnostic Test: Emergence agitation scale
- awake: technique of Anesthesia at the time of airway device removal
  Interventions: Diagnostic Test: Emergence agitation scale
- emergence time (clinical): min: The duration from the time of anesthestic medications stop and the time that patient spontaneously open their eyes
  Interventions: Diagnostic Test: Emergence agitation scale
- Emergence time (entropy): min: time from Entropy value above 60 to 90
  Interventions: Diagnostic Test: Emergence agitation scale

INTERVENTIONS:
Diagnostic Test: Emergence agitation scale — Emergence agitation scale: PAED scale > 10 defined as positive for Emergence agitation (EA) Post hospitalize behavioral questionnaire (PHBQ) positive Post operative behavioral changes defines as 10 % change from sum score of PHBQ
  Other Names: Post operative behavioral changes

SUMMARY:
Emergence agitation (EA) is one of the unpleasant symptoms after general anesthesia. The patient can be irritable, uncooperate, cry, moan and combative behaviors. Sometimes the patient may need to be thrashed to prevent physical harm. The mechanism of EA is still unknown. EA is usually self limiting within 45 to 60 minutes after wake up from anesthesia. The incidence of EA is much higher in pediatric group when compared with adult. In some centre the incidence of EA can be up to 67 % depends on anesthesia technique, race, and child's temperament. Kain et al, reported that the patient who had marked EA tended to have post operative maladaptive behaviors. These maladaptive behaviors such as insomnia, eating disturbance, aggressive behavior and even developmental regression can be happen until one year after anesthesia.

From the previous study, reported that fast emergence was associated with a high incidence of agitation.

This prospective observation study is conducted to determine that emergence time has any effect on EA or not. The authors use process electroencephalogram (entropy) to monitor emergence time which defined as the time which state entropy level over sixty to eighty. Meanwhile, we will evaluate the emergence time by the conventional method which used the time from ceasing anesthesia to the time of eye opening by normal voice stimuli.

The primary outcome of this study is the correlation between emergence time (both from Process EEG and clinical presentation) and incidence of emergence agitation. Two secondary outcomes will be measured. Firstly, the correlation between emergence time and postoperative behavioral changes. Secondly, the relationship between entropy monitoring and clinical symptoms.

ELIGIBILITY:
Inclusion Criteria:

Pediatric patient aged between 3-12 years, ASA physical status I-II who is scheduled for inpatient elective surgery

Exclusion Criteria:

emergency surgery, neurosurgery, antiepileptic medication taken and having ICU admission planning.

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric patient aged between 3-12 years
Sampling Method: Non-Probability Sample
Enrollment: 91 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2013-12 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
emergence agitation | evaluate patient within the first 5 minutes after patient arrive PACU
  Pediatric Anesthesia Emergence delirium scale (PAED) PAED > 10 defined as EA positive

SECONDARY OUTCOMES:
Post operative behavioral changes | up to 7 days postoperative period
  PHBQ (post hospitalization behavioral questionnaires)

CONTACTS AND LOCATIONS:
Overall Officials: Ngamjit Pattaravit, MD, Principal Investigator — Prince of Songkla University
Locations (1):
- Prince of Songkla University, Hat Yai, Changwat Songkhla, Thailand

IPD SHARING:
Plan to Share IPD: Undecided